CLINICAL TRIAL: NCT04455178
Title: The Comparison Between Spironolactone and Indapamide Monotherapy or in Combination With Amlodipine to Reduce the Risk of Heart Failure
Acronym: SIRRHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRRHF
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Hypertension
Keywords: blood pressure; spironolactone
MeSH Terms: conditions — Hypertension | interventions — Spironolactone; Indapamide

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly divided into two groups, taking spironolactone (20mg/tablet) once a day or indapamide (1.5mg/tablet) once a day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Spironolactone 20mg once daily
  Interventions: Drug: Spironolactone
- Indapamide (Active Comparator): Indapamide 1.5mg once daily
  Interventions: Drug: Indapamide

INTERVENTIONS:
Drug: Spironolactone — spironolactone 20mg once daily, up-titrated to 40mg once daily at 4-week or 8-week visit
  Arms: Spironolactone
Drug: Indapamide — indapamide 1.5mg once daily, up-titrated to 3mg once daily at 4-week or 8-week visit
  Arms: Indapamide

SUMMARY:
1. Study name: The comparison between spironolactone and indapamide monotherapy or in combination with amlodipine to reduce thr risk of heart failure (SIRRHF)
2. Medicine: spironolactone (20mg/tablet), indapamide (1.5mg/tablet) and amlodipine (5mg/tablet).
3. Rationale: Our hypothesis of the present trial is that spironolactone is superior to indapamide in cardiovascular prevention in hypertensive patients, with the possible addition of amlodipine. Before a clinical outcome trial is considered, the present feasibility trial is designed to compare the efficacy of antihypertensive regimens based on these two drugs on blood pressure and several measurements of organ damage.
4. Objective: To evaluate the effects of spironolactone (either with or without amlodipine), in comparison with indapamide (either with or without amlodipine), on the extent of blood pressure reduction.
5. Study design: Multi-center (five sites), prospective, randomized, open-label, blinded-end point study with active treatment arm (study duration - 12 weeks)
6. Study population: Men and Women aged over 45 years (n=200) meeting the inclusion/exclusion criteria.
7. Randomization and treatment: After stratification by centers, eligible patients will be randomly divided into two groups, taking spironolactone (20mg tablet) once a day or indapamide (1.5mg tablet) once a day. Spironolactone may be up-titrated to 40mg daily and indapamide may be up-titrated to 3mg daily at 4-week or 8-week visit. At 8-week visit, if needed, we will add amlodipine at 5 or 10 mg once daily.
8. Follow up: 12 weeks.
9. Sample size: a total of 200 patients should be enrolled in the combination.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in June 2020, recruitment will start. Patients enrollment will be performed between June 2020 to November 2020. All patients should be followed up before July 2021.

DETAILED DESCRIPTION:
1. Study name: The comparison between spironolactone and indapamide monotherapy or in combination with amlodipine to reduce thr risk of heart failure (SIRRHF)
2. Medicine: spironolactone (20mg/tablet), indapamide (1.5mg/tablet) and amlodipine (5mg/tablet).
3. Rationale: Our hypothesis of the present trial is that spironolactone is superior to indapamide in cardiovascular prevention in hypertensive patients, with the possible addition of amlodipine. Before a clinical outcome trial is considered, the present feasibility trial is designed to compare the efficacy of antihypertensive regimens based on these two drugs on blood pressure and several measurements of organ damage.
4. Objective: To evaluate the effects of spironolactone (either with or without amlodipine), in comparison with indapamide (either with or without amlodipine), on the extent of blood pressure reduction.
5. Study design: Multi-center (five sites), prospective, randomized, open-label, blinded-end point study with active treatment arm (study duration - 12 weeks)
6. Study population: Men and Women aged over 45 years (n=200) meeting the inclusion/exclusion criteria. Adult subjects with essential hypertension will be included. Specific criteria are as follows:

   Male and female subjects participates (OK with more women is preferred) Age ≥45 years Clinic systolic BP: 140 -179 mmHg (untreated or on monotherapy treatment) Waist Circumference (WC) ≥90 cm for male and ≥85 cm for female
7. Randomization and treatment: After stratification by centers, eligible patients will be randomly divided into two groups, taking spironolactone (20mg tablet) once a day or indapamide (1.5mg tablet) once a day. Spironolactone may be up-titrated to 40mg daily and indapamide may be up-titrated to 3mg daily at 4-week or 8-week visit. At 8-week visit, if needed, we will add amlodipine at 5 or 10 mg once daily.
8. Follow up: 12 weeks. Patients will be followed up every 4 weeks. Ambulatory and office blood pressure will be measured. Medical history should be recorded. Clinical examinations including blood biochemical tests (serum creatinine, uric acid and electrolytes) should be performed.
9. Sample size: a total of 200 patients should be enrolled in the combination.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in June 2020, recruitment will start. Patients enrollment will be performed between June 2020 to November 2020. All patients should be followed up before July 2021.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China

ELIGIBILITY:
Inclusion Criteria:

Adult subjects with essential hypertension will be included. Specific criteria are as follows

1. Male and post menopause female subjects participates (OK with more women is preferred)
2. Age ≥45 years
3. Clinic systolic BP: 140 -179 mmHg (untreated or on monotherapy treatment)
4. Waist Circumference (WC) ≥90 cm for male and ≥85 cm for female

Exclusion Criteria:

1. Confirmed secondary hypertension
2. Hyperkalemia (serum potassium concentration ≥5.0 mmol/L) or hypokalemia (serum potassium concentration ≤3.5 mmol/L)
3. Contraindication for the treatment drugs or current use of spironolactone, indapamide or amlodipine
4. Chronic kidney disease (eGFR≤45 ml/min 1.73 m² or serum creatinine ≥ 2 mg/dl)
5. Expected lifespan ≤6 months
6. Treated subjects in whom withdrawal of antihypertensive treatment is deemed unethical by the investigator (e.g. because of the existence of compelling indications other than hypertension for continuous use of previously used antihypertensive agent)
7. Contraindications to study treatments as detailed in the relative Summaries of medical Product Characteristics for spironolactone, indapamide or amlodipine (this includes hypersensitivity, pregnancy and lactation)
8. Diagnosed cardiovascular diseases other than hypertension (coronary heart disease, heart failure or left ventricular systolic dysfunction of any degree, atrial fibrillation or frequent arrhythmias, valvular or congenital heart disease, cardiomyopathies, cerebrovascular disease, peripheral artery disease, or aortic aneurysm)
9. Subjects with conditions other than those mentioned above, where compelling indications for the use of any specific class of antihypertensive medication exist, according to the current (e.g. European Society of Cardiology) guidelines
10. Other conditions deemed relevant by the investigator (including respiratory disorders, liver disease, renal disease, thyroid disorders)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
pulse wave velocity | 12 weeks

SECONDARY OUTCOMES:
systolic blood pressure | 12 weeks

OTHER OUTCOMES:
NT-proBNP | 12 weeks
  NT-proBNP level will be measured by Roche Diagnostics.
Type I & III procollagen | 12 weeks
  Type I & III procollagen level will be measured using a commercial ELISA kit

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Dongtai Renmin Hospital, Dongtai, Jiangsu
  - Kunshan First Renmin Hospital, Kunshan, Jiangsu
  - Changzhi Heping Hospital, Changzhi, Shanxi
  - Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai